CLINICAL TRIAL: NCT02141724
Title: Assessment of Wheelchair Positioning and Pain in Adults Patients With Neuromuscular Disorder
Brief Title: Wheelchair Positioning and Pain in Neuromuscular Patients
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Fondation Garches (Other); Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 0946927B
Record Dates: First submitted 2014-05-13; First posted 2014-05-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Adult Patients With Neuromuscular Disorders Using Wheelchair
Keywords: Neuromuscular; Wheelchair; Pain; Bedsore; Trouble postural
MeSH Terms: conditions — Pain; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- neuromuscular patients: neuromuscular patients using wheelchair
  Interventions: Other: Positioning consultation

INTERVENTIONS:
Other: Positioning consultation — Assessment of pain,bedsores and postural troubles

SUMMARY:
A retrospective study with the patients having a positioning consultation at hospital, between 2009 and 2014. In every neuromuscular disorder, the investigators describe the population seen in consultation, the aim of consultation, the postural problem observed in wheelchair, pain when sitting in wheelchair, and pressure ulcer.

DETAILED DESCRIPTION:
Postural problem is described with MCPAA (Measure of Postural Control in Sitting Position, created by B. GAGNON, physiotherapist in Quebec) : we look at pelvic obliquity, pelvic rotation, pelvic anteversion or retroversion, trunk slope and rotation, kyphotic or scoliotic posture, neck posture and legs posture. We evaluate if these deformities are soft, moderate or severe, and if they are relievable

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with neuromuscular disorder
* using wheelchair
* Patient having a positioning consultation in GARCHES Hospital

Exclusion Criteria:

* refusal to participate to the protocol
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with neuromuscular disordres using wheelchair.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Postural disorders | 2h

SECONDARY OUTCOMES:
Number of patient with Pain | 15 minutes

OTHER OUTCOMES:
Bedsores | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: PELLEGRINI Nadine, MD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France